CLINICAL TRIAL: NCT01820390
Title: Optimizing DBS Electrode Placement and Programming Using a Combination of High-Field MRI, Intraoperative Electrophysiology, and Computational Modeling.
Brief Title: Optimizing DBS Electrode Placement and Programming
Status: Withdrawn | Type: Observational
Why Stopped: Funding discontinued.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-1837
Record Dates: First submitted 2013-01-14; First posted 2013-03-28 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease; Essential Tremor
Keywords: Deep Brain Stimulation (DBS); Parkinson's Disease; Essential Tremor
MeSH Terms: conditions — Parkinson Disease; Essential Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Deep brain stimulation (DBS) has become the primary surgical therapy for the treatment of motor symptoms associated with Parkinson's disease (PD), and for essential tremor (ET). Although an effective and relatively safe procedure with expanding indications, opportunities exist for the optimization of the current procedure.

The investigators therefore propose, in a group of patients undergoing DBS surgery for the treatment of PD or ET, to use a combination of high-field imaging modalities, intraoperative electrophysiology, external sensor interfaces, and computational modeling, to gather information on the utility of using these techniques to optimize DBS electrode placement and programming.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of idiopathic Parkinson's disease or essential tremor
* Ability to provide informed consent

Exclusion Criteria:

* Claustrophobia or other conditions that prevent undergoing MR imaging
* MMSE score < 23
* Significant neurological diagnosis other than PD or ET.
* Idiopathic dystonia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the population of patients undergoing DBS surgery at the University of Minnesota Medical Center, for the treatment of (1) Parkinson's disease, or (2) essential tremor.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Distance between Electrophysiology Results and Modeling Predictions (mm) | 1 week
  A comparison between electrophysiology results and modeling predictions will be made post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Aviva D Abosch, M.D., Ph.D., Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Department of Neurosurgery, University of Colorado, Aurora, Colorado
  - University of Colorado, Aurora, Colorado

REFERENCES:
- [Background] Abosch A, Lanctin D, Onaran I, Eberly L, Spaniol M, Ince NF. Long-term recordings of local field potentials from implanted deep brain stimulation electrodes. Neurosurgery. 2012 Oct;71(4):804-14. doi: 10.1227/NEU.0b013e3182676b91. PMID 22791039
- [Background] Duchin Y, Abosch A, Yacoub E, Sapiro G, Harel N. Feasibility of using ultra-high field (7 T) MRI for clinical surgical targeting. PLoS One. 2012;7(5):e37328. doi: 10.1371/journal.pone.0037328. Epub 2012 May 17. PMID 22615980
- [Background] Lenglet C, Abosch A, Yacoub E, De Martino F, Sapiro G, Harel N. Comprehensive in vivo mapping of the human basal ganglia and thalamic connectome in individuals using 7T MRI. PLoS One. 2012;7(1):e29153. doi: 10.1371/journal.pone.0029153. Epub 2012 Jan 3. PMID 22235267
- [Background] Ince NF, Gupte A, Wichmann T, Ashe J, Henry T, Bebler M, Eberly L, Abosch A. Selection of optimal programming contacts based on local field potential recordings from subthalamic nucleus in patients with Parkinson's disease. Neurosurgery. 2010 Aug;67(2):390-7. doi: 10.1227/01.NEU.0000372091.64824.63. PMID 20644424